CLINICAL TRIAL: NCT07150793
Title: Real-world Treatment and Burden of Chronic Myeloid Leukemia Patients in Japan - A Retrospective Claims Database Analysis
Brief Title: A Study of Real-world Treatment and Burden of Chronic Myeloid Leukemia Patients in Japan
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107AJP11
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: Tyrosine Kinase Inhibitor; Real-world
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- CML Cohort: Patients diagnosed with chronic phase CML who received treatment with a TKI in Japan between 01 January 2011 and 31 December 2019.

SUMMARY:
The main goal of this study was to describe treatment patterns of patients with chronic myeloid leukemia (CML) who were treated with tyrosine kinase inhibitors (TKIs) in Japan.

This was a retrospective observational study with secondary use of data from the Medical Data Vision (MDV) hospital-based database. The index date was the date of the first prescription of any TKI of interest registered within the selection period (01 January 2011 to 31 December 2019). The follow-up period was from the index date until the end of the study period, end of continuous follow-up in the MDV database, or death, whichever came first.

ELIGIBILITY:
Patients who met all the below inclusion criteria and none of the exclusion criteria were included in the study.

Inclusion criteria:

* Patients who had at least one TKI prescription during the selection period,
* a confirmed diagnosis of chronic phase CML recorded before or at the index date,
* were aged 15 years or older at the index date, and
* had at least 12-months continuous pre-index period.

Exclusion criteria:

* Patients who had at least one TKI prescription in the 12 months preceding the index date (washout period to catch the 1st line of treatment [LoT]),
* a confirmed diagnosis of CML blast crisis or accelerated phase recorded prior to, at, or within 6 months after the index date,
* a confirmed diagnosis of acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) within 6 months after the index date,
* a medical record of chemotherapy (not including hydroxyurea) within 6 months after the index date,
* a stem cell transplant procedure recorded during the pre-index period.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Number of Patients by Line of Treatment (LoT) and TKI Received | Up to approximately 9 years
  TKIs included imatinib, bosutinib, dasatinib, nilotinib, and ponatinib.
Number of Patients who Switched TKI Treatment by LoT and TKI | Up to approximately 9 years
  TKIs included imatinib, bosutinib, dasatinib, nilotinib, and ponatinib.
Number of Patients who Discontinued TKI Treatment by Type of TKI | Up to approximately 9 years
  TKIs included imatinib, bosutinib, dasatinib, nilotinib, and ponatinib.
Number of Patients who Discontinued TKI Treatment for at Least One Year by Type of TKI | Up to approximately 9 years
  TKIs included imatinib, bosutinib, dasatinib, nilotinib, and ponatinib.
Number of Patients who Restarted any TKI Treatment After Discontinuing the TKI of Interest by Type of TKI | Up to approximately 9 years
  TKIs included imatinib, bosutinib, dasatinib, nilotinib, and ponatinib.
TKI Dose by LoT | Baseline, up to approximately 9 years
  TKIs included imatinib, bosutinib, dasatinib, nilotinib, and ponatinib.
TKI Persistence Rate by LoT | Months 6, 12, 18, and Year 5
Duration of TKI Treatment by LoT | Up to approximately 9 years

SECONDARY OUTCOMES:
Annual Incidence of Inpatient and Outpatient Visits by LoT | Up to approximately 9 years
Annual Mean Cost of All-cause Healthcare Resource Use by LoT | Up to approximately 9 years
  All-cause care included inpatient and outpatient visits. The following costs were calculated in Japanese yen (JPN):
  * Total costs
  * Inpatient costs
  * Outpatient costs
  * Pharmacy costs
Annual Incidence of CML-related Healthcare Resource Use by LoT | Up to approximately 9 years
  CML-related care included:
  * Major BCR-ABL1 procedures (diagnostic and response to treatment testing)
  * Complete blood count testing - peripheral blood general testing
  * Hematological examination diagnosis fee
  * TKI prescriptions
Annual Mean Cost of CML-related Healthcare Resource Use by LoT | Up to approximately 9 years
  CML-related care costs were calculated in Japanese Yen (JPY) and included the following:
  * Total CML-related costs
  * Major BCR-ABL1 procedure costs
  * Complete blood count testing - peripheral blood general testing costs
  * Hematological examination costs
  * TKI prescription costs
Number of Patients With Adverse Events by TKI | Up to approximately 9 years
  TKIs included imatinib, bosutinib, dasatinib, nilotinib, and ponatinib.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States